CLINICAL TRIAL: NCT07321223
Title: Comparison of Different Doses of Vitamin D Supplementation on Glycated Haemoglobin and Blood Glucose Parameters With Type II Diabetes Mellitus Having Vitamin d Deficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/880/2021
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Diabetes (DM); Vitamin D Deficiency
Keywords: Diabetes Mellitus; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group-1 (Experimental): Treatment vitamin D capsules with different dosage (50,000IU) once a week for 90days
  Interventions: Dietary Supplement: Vitamin D
- Placebo (No Intervention): Only Metformin and Balance Diet
- Treatment Group 2 (Experimental): Treatment vitamin D capsules with different dosage (200000IU) once a week for 90days
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D supplement capsules (50,000 IU, 200000 IU)
  Arms: Treatment Group 2; Treatment Group-1

SUMMARY:
COMPARISON OF DIFFERENT DOSES OF VITAMIN D SUPPLEMENTATION ON GLYCATED HEMOGLOBIN (HbA1c) and BLOOD GLUCOSE PARAMETRS IN PATIENTS WITH TYPE 2 DIABETES MELLITUS HAVING VITAMIN D DEFICIENCY"

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed of T2DM with the age of 40-70 years from both genders taking only metformin with an Hb1Ac range of 7.5-9% and 25-hydroxy Vitamin D levels (25[OH]D) <20ng/ml. Exclusion Criteria: Individuals

Exclusion Criteria: Individuals with the following conditions will not be included as participants;

* Inability or unwilling to participate or Clinical proximal myopathy
* Renal, hepatic, endocrinological disorders or malignancies on basis of history
* Serum calcium levels > 10.5mg/dl
* Use of insulin or any change in dosage of current hypoglycemic medications during last 3 months
* Intake of vitamin D, calcium or omega 3 supplements within the past 3 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 90 days

SECONDARY OUTCOMES:
Blood Safety Profile (LFTs, RFTs) | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- PAF Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes